CLINICAL TRIAL: NCT04246567
Title: Evaluation of the Effect of Sevoflurane and Propofol Hypotensive Anesthesia on Blood Antioxidant Levels and HIF 1 Levels
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Ethics approval is expected from the pharmaceutical institution for the study which has received the local ethics committee approval.
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Ayse02
Record Dates: First submitted 2020-01-22; First posted 2020-01-29 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Hypoxemia During Surgery; Hypoxia
Keywords: hypotensive anesthesia; HIF 1a; total intravenous anesthesia; inhalation anesthesia
MeSH Terms: conditions — Hypoxia | interventions — Arterial Pressure; Fentanyl

STUDY DESIGN:
Intervention Model Description: A total of 60 ASA 1 patients aged between 18-55 who underwent elective rhinoplasty surgery were included the study.The patients were divided into two groups. One group received hypotensive anesthesia with total intravenous anesthesia technique according to MBP and the other group received hypotensive anesthesia with inhalation anesthesia technique. Blood samples were taken from all patients before anesthesia induction and 30. ,60. ,120. second of intraoperative period for TAS, TOS, HIF 1a. At the and of the operation patients were fallowed in the post anesthesia care unit for 30 minutes and pain and nause vomiting scores were evaluated. İn addition, surgical satisfaction and bleeding scores and anesthetic consumption of both groups were recorded
Who Masked: Participant
Masking Description: The investigators divided the patients to two groups. Patients were divided into two groups with a lottery. Surgeons did not know which hypotensive anesthesia technique were used. And surgeons evaluated surgical satisfaction and bleeding scores
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total intravenous anesthesia technique for group 1 patients (Active Comparator): Procedure/Surgery:Mean Blood Pressure (MBP) Mean blood pressure (MBP) 50-65 mmHg was applied with 6-10 mg / kg / h propofol and 0.0,4mcg / kg remifentanyl infusion / min. When BIS values are between 40-60 and muscle relaxation was sufficient (TOF 0), a 20% increase in the initial blood pressure and heart rate values of patients were added to 0.5 mcg / kg fentanyl. All patients received 5-8 ml / kg / h IV infusion of balanced electrolyte solution (Isolyte-S) during the operation.
  Hemodynamic parameters (HR, SBP, OCD), BIS,TOF and SpO2 were recorded at 5 minute intervals.
  Blood samples were taken from patients during preop preparation (t0), 30th minute (t1), 1st hour (t2) and 2nd hour (t3) of the operation. 5 ml of blood was taken from the untreated arm of all patients to the HIF1a, TAS and TOS values and sent to the biochemistry laboratory
  Interventions: Procedure: Mean Blood Pressure (MBP); Drug: Add to 0.5 mcg / kg fentanyl.
- Inhalation anesthesia technique for group 2 patients (Active Comparator): Procedure/Surgery:Mean Blood Pressure (MBP) Mean blood pressure (MBP) 50-65 mmHg was applied with 40% Oxygen 60% N2O2 and Sevoflurane at a concentration of 1.5-3.5% with 2 L / minTGA to provide a value of BIS between 40-60. When BIS values are between 40-60 and muscle relaxation was sufficient (TOF 0), a 20% increase in the initial blood pressure and heart rate values of patients were added to 0.5 mcg / kg fentanyl. All patients received 5-8 ml / kg / h IV infusion of balanced electrolyte solution (Isolyte-S) during the operation.
  Hemodynamic parameters (HR, SBP, OCD), BIS,TOF and SpO2 were recorded at 5 minute intervals.
  Blood samples were taken from patients during preop preparation (t0), 30th minute (t1), 1st hour (t2) and 2nd hour (t3) of the operation. 5 ml of blood was taken from the untreated arm of all patients to the HIF1a, TAS and TOS values and sent to the biochemistry laboratory
  Interventions: Procedure: Mean Blood Pressure (MBP); Drug: Add to 0.5 mcg / kg fentanyl.

INTERVENTIONS:
Procedure: Mean Blood Pressure (MBP) — Mean blood pressure (MBP) for patients 50-65 mmHg
Drug: Add to 0.5 mcg / kg fentanyl. — When BIS values are between 40-60 and muscle relaxation was sufficient (TOF 0), a 20% increase in the initial blood pressure and heart rate values of patients were added to 0.5 mcg / kg fentanyl.

SUMMARY:
The aim of this study to evaluate the patients who underwent controlled hypotensive anesthesia under standardized depth of anesthesia with total intravenous anesthesia or inhalation anesthesia; preoperative and 30. ,60. ,120. second of intraoperative period blood HIF 1a, TAS, TOS measurement and to investigate tissue hypoxia secondary to hypotensive anesthesia and the changes of the mediators at the tissue level and which hypotensive anesthesia technique is related.

DETAILED DESCRIPTION:
Controlled hypotension is the voluntary reversible reduction of arterial blood pressure. Hypotensive anesthesia is a method of anesthesia in which blood pressure is reduced in a controlled manner, especially in certain surgeries. İt reduces intraoperative bleeding and need for blood transfusion and provides a clean surgical vision in narrow-field surgeries or with high bleeding potential. Hypotensive anesthesia can be performed according to mean blood pressure (MBP) or systolic blood pressure (SBP).

A non-invasive cerebral oximeter is used to see the changes in the brain due to high oxygen-dependent metabolism during induction and maintenance of anesthesia.

Hypoxia inducible factor (HIF) is a transcription factor involved in cell adaptation mechanism activated in response to hypoxia.

The biological activity of HIF 1 is determined by the expression and activity of the HIF 1a subunit.

Total antioxidant status (TAS) shows the total effect of all antioxidants in the human body and total oxidant status (TOS) shows the total effect of oxidants.

Near Infrared Spectroscopy (NIRS) allows continuous and non-invasive monitoring of cerebral oxygenation. HIF 1a, TAS and TOS are laboratory markers that predict tissue oxygenation and perfusion.

Hypotensive anesthesia can be performed according to both MBP and SBP. However, in our study that follow-up MBP is more advantageous/protective, although it is not supported by very strong data. The investigators recommend hypotensive anesthesia compared to MBP; but further studies are needed

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old
* ASA Physical Status Classification System 1
* Undergoing to Elective rhinoplasty

Exclusion Criteria:

* Patients have any autoimmune disease
* Smoking of patients
* Development of any allergic reaction during the procedure
* Failure to collect blood to be examined at the appropriate time
* Body mass index is less than 19 or greater than 30

Termination criteria

* Development of severe hypotension and bradycardia during measurements
* Development of severe drug allergy during follow-up
* In the event of any complications related to the surgical procedure

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the relationship between hypotensive anesthesia technique and tissue hypoxia by HIF1a | Change from Baseline HIF 1a 30th minute (t1), 1st hour (t2) and 2st hour (t3)
  Under normoxic conditions, HIF 1a protein can hardly be detected, but when hypoxia starts, its expression starts within 2 minutes and peaks at 4-8 hours of hypoxia.
  5 ml blood was taken into MiniCollect® tubes from the venous cannula placed before anesthesia (t0) induction for measure HIF 1a,TAS and TOS. 30th minute (t1), 1st hour (t2) and 2nd hour (t3) of the operation 5 ml of blood was taken again from the untreated arm of all patients to the HIF1a, TAS and TOS values and sent to the biochemistry laboratory. The collected blood was centrifuged at 2000 x g for 10 minutes and the separated sera were sent to the biochemical laboratory to be stored at -80 ° C until the study was performed.
Evaluation of the relationship between hypotensive anesthesia technique and tissue hypoxia by the concentration of TAS | Change from Baseline TAS levels at 30th minute (t1), 1st hour (t2) and 2st hour (t3)
  Plasma TAS and TOS levels are measured with a commercial kit developed by Erel. Values for plasma TAS are expressed in millimeters by the Trolox value per liter.
  5 ml blood was taken into MiniCollect® tubes from the venous cannula placed before anesthesia (t0) induction for measure HIF 1a,TAS and TOS. 30th minute (t1), 1st hour (t2) and 2nd hour (t3) of the operation 5 ml of blood was taken again from the untreated arm of all patients to the HIF1a, TAS and TOS values and sent to the biochemistry laboratory. The collected blood was centrifuged at 2000 x g for 10 minutes and the separated sera were sent to the biochemical laboratory to be stored at -80 ° C until the study was performed.
Evaluation of the relationship between hypotensive anesthesia technique and tissue hypoxia by the concentration of TOS | Change from Baseline TOS levels at 30th minute (t1), 1st hour (t2) and 2st hour (t3)
  Measurement for TOS is calibrated with hydrogen peroxide and the results are expressed in micromolar by the hydrogen peroxide value per liter (mmol H2O2 equiv / L).5 ml blood was taken into MiniCollect® tubes from the venous cannula placed before anesthesia (t0) induction for measure HIF 1a,TAS and TOS. 30th minute (t1), 1st hour (t2) and 2nd hour (t3) of the operation 5 ml of blood was taken again from the untreated arm of all patients to the HIF1a, TAS and TOS values and sent to the biochemistry laboratory. The collected blood was centrifuged at 2000 x g for 10 minutes and the separated sera were sent to the biochemical laboratory to be stored at -80 ° C until the study was performed.

SECONDARY OUTCOMES:
surgical satisfaction | postoperative 1 minute
  At the end of the surgery surgeons evaluated surgical satisfaction. the investigators used surgeon satisfaction score which one is performing like that 1- bad 2-moderate 3-good 4-excellent
bleeding scores | postoperative 1 minute
  At the end of the surgery surgeons evaluated bleeding scores. the investigators used bleeding score which one is performing like that 0-No bleeding 1-minor bleeding no aspiration required 2- Minor bleeding, aspiration required 3-minor bleeding, frequent aspiration required, 4-Moderate bleeding, visible only with aspiration 5- Severe bleeding, frequent aspiration required and very hard to perform surgery
anesthetic consumption for group 1 propofol consumption (mg) and remifentanyl consumption(microgram) | postoperative 1 minute
  Standard anesthesia induction and propofol and remifentanil infusion were applied to group 1 patients with TIVA technique.
  Standard anesthesia induction and 40% Oxygen 60% N2O2 and Sevoflurane at a concentration of 1.5-3.5% with 2 L / minTGA were applied to group 2 patients with inhalation anesthesia technique
anesthetic consumption for group 2 N2O2 consumption (ml) and sevoflurane consumption (ml) | postoperative 1 minute
  Standard anesthesia induction and 40% Oxygen 60% N2O2 and Sevoflurane at a concentration of 1.5-3.5% with 2 L / minTGA were applied to group 2 patients with inhalation anesthesia technique

CONTACTS AND LOCATIONS:
Overall Officials: Hayrettin Daşkaya, MD, Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)